CLINICAL TRIAL: NCT01218074
Title: Platelets Antiaggregation Control Enhancement Study: an Independent Randomized Blind Prospective Study
Brief Title: Platelets Antiaggregation Control Enhancement (PACE) Study
Acronym: PACE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Principal Investigator, Luca Weltert, Project Leader Luca Weltert, Cardiochirurgia E.H.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00-04
Record Dates: First submitted 2010-10-05; First posted 2010-10-11 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Bleeding; Blood Transfusion
Keywords: bleeding; blood sparing procedure; desmopressin; aggregometry; thromboelastography
MeSH Terms: conditions — Hemorrhage | interventions — Thrombelastography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thromboelastography alone (Active Comparator): Patients undergo standard of care Thromboelastography to evaluate overall coagulation performances.
  Interventions: Device: Thromboelastography Alone
- Aggregometry+Tromboelastography (Experimental): Patients undergo standard thromboelastography and subsequent aggregometry to test effectiveness of residual antiaggregation drugs. Patients found to have altered value undergo optimization with desmopressin.
  Interventions: Device: Aggregometry+Thromboelastography

INTERVENTIONS:
Device: Aggregometry+Thromboelastography — Patients undergo standard thromboelastography and subsequent aggregometry to test effectiveness of residual antiaggregation drugs. Patients found to have altered value undergo optimization with desmopressin.
  Arms: Aggregometry+Tromboelastography
Device: Thromboelastography Alone — Patients undergo standard of care Thromboelastography to evaluate overall coagulation performance.
  Arms: Thromboelastography alone

SUMMARY:
Many patients undergo cardiac surgery without proper suspension of antiaggregation drugs. This is blamed to increase dramatically bleeding and use of allogenic blood transfusions. The investigators test the hypothesis that routine use of aggregometry could show antiaggregated patient and lead to normalization of platelet function via administration of Desmopressin thus limiting bleeding and transfusions.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing surgical myocardial revascularization.

Exclusion Criteria:

* none.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-12; Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Bleeding Volume | 12 hours after end of operation
  Total amount of bleeding in the first 12 hours after cardiac surgery expressed as milliliters of blood in the chest drains reservoir.

SECONDARY OUTCOMES:
Use of allogenic blood transfusions. | In hospital stay (usually 5 to 8 days after operation)
  Number of allogenic blood units transfused per patients during the full hospital stay, usually 5 to 8 days after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- European Hospital, Rome, Italy